CLINICAL TRIAL: NCT05741632
Title: Safety Profile Comparison of Undiluted Intracameral Moxifloxacin vs. Levofloxacin in Cataract Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Ferron Par Pharmaceuticals (Unknown)
Responsible Party: Principal Investigator, Arcci Pradessatama, Ophthalmology Department Resident, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-10-1262; KET-1303/UN2.F1/ETIK/PPM.00.02 (Other: Komite Etik Penelitian Kesehatan FKUI)
Record Dates: First submitted 2023-02-14; First posted 2023-02-23 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Cataract
Keywords: Moxifloxacin; Levofloxacin; Cataract surgery
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Intervention Model Description: First group will receive Moxifloxacin intracameral during surgery Second group will receive Levofloxacin intracameral during surgery
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participant will be masked receiving treatment, post operative eye drops of both arms is the same. Subject allocation is blinded to investigator and outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moxifloxacin (Experimental): Subjects will receive 0.1 cc undiluted non preserved intracameral Moxifloxacin during cataract surgery.
  Interventions: Drug: Moxifloxacin Ophthalmic Solution
- Levofloxacin (Active Comparator): Subjects will receive 0.1 cc undiluted non preserved intracameral Levofloxacin during cataract surgery.
  Interventions: Drug: Levofloxacin Ophthalmic

INTERVENTIONS:
Drug: Moxifloxacin Ophthalmic Solution — Moxifloxacin solution 0.1 cc undiluted, self preserved, injected into intracamera at the end of cataract surgery
  Other Names: Molcin(R)
  Arms: Moxifloxacin
Drug: Levofloxacin Ophthalmic — Levofloxacin solution 0.1 cc undiluted, self preserved, injected into intracamera at the end of cataract surgery
  Other Names: Cravit(R)
  Arms: Levofloxacin

SUMMARY:
The goal of this randomized clinical trial study is to compare safety profile undiluted intracameral moxifloxacin vs levofloxacin during cataract surgery. The main question it aims to answer is whether moxifloxacin and levofloxacin have similar safety profile.

Participant will be randomized into two treatment arms. All participant will receive standardized treatment before, during, and after surgery and will be followed up at one day, one week, and one month after surgery.

DETAILED DESCRIPTION:
This study aims to observe the safety profile in patient receiving cataract surgery who receives moxifloxacin and levofloxacin intracamerally during the surgery. Safety profile defined as visual acuity, intraocular pressure, corneal endothelial cell density, central corneal thickness, anterior chamber reactions, and central macular thickness. Parameters are obtained before the surgery, 1 day, 1 week, and 1 month after surgery. Subjects are randomized to two treatment arms: (1) receiving undiluted moxifloxacin 0.1 cc during surgery; (2) receiving undiluted levofloxacin 0.1 cc during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Immature senile cataract in one or both eye
* Agree to be included and signed informed consent

Exclusion Criteria:

* Have a history of allergy to moxifloxacin or levofloxacin or any other antibiotics
* Other ocular comorbid such as uveitis, glaucoma, diabetic retinopathy, pseudoexfoliation, and endothelial disorders
* Ocular surgery prior to study
* Sign of infection or inflammation around the eye
* Cataract density more than grade 4 according to Lens Opacities Classification System (LOCS) III grading
* Corneal endothelial cell density < 1500 cell/ mm2
* Anterior chamber depth < 2.5 mm
* Diabetes mellitus type 2

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
Endothelial cell density | 1 month
  Corneal endothelial cell density measured using specular microscopy

SECONDARY OUTCOMES:
Central corneal thickness | 1 month
  Central corneal thickness (in nm) measured using specular microscopy
Central macular thickness | 1 month
  Central macular thickness (in nm) measure using optical coherence tomography
Anterior chamber cell reactions | 1 month
  Anterior chamber cell reactions measured in Standardization of Uveitis Nomenclature (SUN) grading. Values consist of 0, trace, 1+, 2+, 3+, and 4+. Higher grading score means more inflammatory reaction which is worse.
Intraocular pressure | 1 month
  Intraocular pressure (in mmHg) measured using automated non contact tonometer

CONTACTS AND LOCATIONS:
Overall Officials: Arcci Pradessatama, MD, Principal Investigator — RSCM Kirana
Locations (1):
- Fakultas Kedokteran Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Melega MV, Alves M, Cavalcanti Lira RP, Cardoso da Silva I, Ferreira BG, Assis Filho HL, Pedreira Chaves FR, Martini AAF, Dias Freire LM, Reis RD, Leite Arieta CE. Safety and efficacy of intracameral moxifloxacin for prevention of post-cataract endophthalmitis: Randomized controlled clinical trial. J Cataract Refract Surg. 2019 Mar;45(3):343-350. doi: 10.1016/j.jcrs.2018.10.044. Epub 2019 Jan 25. PMID 30691922
- [Background] Chang DF, Prajna NV, Szczotka-Flynn LB, Benetz BA, Lass JH, O'Brien RC, Menegay HJ, Gardner S, Shekar M, Rajendrababu S, Rhee DJ. Comparative corneal endothelial cell toxicity of differing intracameral moxifloxacin doses after phacoemulsification. J Cataract Refract Surg. 2020 Mar;46(3):355-359. doi: 10.1097/j.jcrs.0000000000000064. PMID 32050222
- [Background] Lucena NP, Pereira IMS, Gaete MIL, Ferreira KSA, Melega MV, Lira RPC. Intracameral moxifloxacin after cataract surgery: a prospective study. Arq Bras Oftalmol. 2018 Apr;81(2):92-94. doi: 10.5935/0004-2749.20180022. PMID 29846429